CLINICAL TRIAL: NCT02434874
Title: Randomized, Multi-Center Pivotal Study for Sacral Nerve Stimulation to Treat Refractory Urgency Urinary Incontinence With Wireless Neuromodulation Technology
Brief Title: Sacral Nerve Stimulation to Treat Urgency Urinary Incontinence With Wireless Neuromodulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study will no longer take place, the study did not begin or accrue subjects.
Sponsor: Uro Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-00780
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Urinary Incontinence, Urge
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Immediate Activation (Experimental): Subjects randomized to this group will have the StimGuard Sacral Nerve Stimulator System activated immediately.
  Interventions: Device: StimGuard Sacral Nerve Stimulator System
- Delayed Activation (Other): Subjects randomized to this group will have the StimGuard Sacral Nerve Stimulator System activated after 90 days.
  Interventions: Device: StimGuard Sacral Nerve Stimulator System

INTERVENTIONS:
Device: StimGuard Sacral Nerve Stimulator System — The StimGuard Sacral Nerve Stimulator System is a wirelessly powered neurostimulator for urge urinary incontinence. This technology includes a quadripolar stimulator with an embedded receiver. The energy source is a small, external, rechargeable transmitter, which is worn by the patient. The transmitter sends the therapy program and power through the skin and to the receiver.

SUMMARY:
The purpose of this pivotal study is to illustrate the safety and effectiveness of the StimGuard Sacral Nerve Stimulation (SNS) System in the treatment refractory urge incontinence. This is a prospective, randomized, controlled, multi-center, study in which 92 subjects will receive a StimGuard SNS System.

DETAILED DESCRIPTION:
The StimGuard SNS System is utilized for the treatment of refractory urgency urinary incontinence as defined by the International Continence Society (ICS) Standardization of Terminology Committees Joint Report as the observation of involuntary leakage from the urethra synchronous with the sensation of a sudden, compelling desire to void that is difficult to defer. The system provides treatment by delivering small controlled electrical pulses to the sacral nerves, as these nerves have been shown to regulate the micturition cycle.

In this study, subjects will be randomized into one of two groups with a 1:1 ratio after enrollment. Subjects will either be randomized to an immediate or a delayed activation group. An intraoperative test will be performed, and all subjects will receive a permanent implant if they have an appropriate motor nerve root response without significant discomfort at 5 mA amplitude or less.

ELIGIBILITY:
Inclusion Criteria:

A. Diagnosis of overactive bladder with urgency urinary incontinence; B. Women and men ≥ 18 years of age; C. At least 4 incontinent episodes associated with urge on a 3 day voiding diary with at least 1 each 24 hour day; D. Self-reported bladder symptoms present > 6 months; E. Self-reported failed conservative care > 6 months (i.e., pharmacology, dietary restriction, fluid restriction, bladder training, behavioral modification, pelvic muscle training, biofeedback, etc.); F. Off all antimuscarinics and beta-3 adrenergic agonists for at least 2 weeks prior to enrollment; G. Have no reported history of urethral obstruction/stricture, bladder calculi or bladder tumor; H. Normal upper urinary tract function; I. Capable of giving informed consent; J. Capable and willing to follow all study related procedures.

Exclusion Criteria:

A. Any active implantable electronic device regardless of whether stimulation is ON or OFF; B. Pregnant as confirmed by a urine pregnancy test or plan to become pregnant during the following 12 months period; C. Less than 1 year post partum and/or are breast-feeding; D. Neurogenic bladder; E. Botox use in bladder or pelvic floor muscles in the past six months; F. Taking alpha-blocker therapy; G. Have a PVR >150 cc at baseline; H. Primary complaint of stress urinary incontinence; I. Current urinary tract infection (UTI); J. Previous treatment with sacral neuromodulation; K. Previous treatment with tibial nerve stimulation, pelvic floor muscle stimulation, or biofeedback within the past 60 days; L. Conditions requiring Magnetic Resonance Imaging (MRI) evaluation or diathermy procedures; M. Inability to operate the StimGuard SNS System; N. Diabetes with peripheral nerve involvement or have severe uncontrolled diabetes (HbA1C 8.5 or greater); O. History of coagulopathy or bleeding disorder; P. History of pelvic pain as primary diagnosis (VAS score of > 4); Q. Anatomical restrictions such that device placement is not possible; R. Currently participating or have participated within the past 30 days in any clinical investigation involving or impacting urinary or renal function; S. Life expectancy of less than 5 years; T. Inability to independently comprehend and complete the questionnaires and diaries; U. Unsuitable for enrollment in study by the investigators based on subjects' history or physical examination (including bleeding disorders or anticoagulant medications, and peripheral neuropathy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in number of urge related incontinence episodes | 3 Months
  Self reported on a 3-day voiding diary
Incidence and severity of adverse events | Up to 12 months

SECONDARY OUTCOMES:
Proportion of subjects with a reduction in the degree of urgency as measured by PPIUS | 3 Months
  Self reported on a 3-day voiding diary
Proportion of subjects with a reduction in the number of voids compared to baseline | 3 Months
  Self reported on a 3-day voiding diary
Improved quality of life function via the Incontinence Quality of Life Scale (I-QOL) | 3 Months
  Quesionnaire

OTHER OUTCOMES:
Proportion of subjects dry | 12 months
  Self reported on a 3-day voiding diary
Number of Episodes associated with urge | 12 months
  Self reported on a 3-day voiding diary
Proportion of subjects reporting improvement | 12 Months
  Measured by Global Response Assessment as "moderately" or "markedly improved"
Improved quality of life function via Overactive Bladder Questionnaire (OAB-Q) | 12 Months
  Questionnaire
Improved quality of life function via Idiopathic Overactive Bladder Symptom Score (iOABSS) | 12 Months
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Beaumont Hospital, Royal Oak, Michigan, United States